CLINICAL TRIAL: NCT02590991
Title: A Follow-up Clinical Study to Investigate the Long Term Effect of Supplementation of Pre- and Probiotics in Early Life in Children Born by Caesarean Section (Julius SN Follow-up 1)
Brief Title: Follow-up Study to Investigate Long Term Effect of Supplementing Pre- and Probiotics in Children Born by C-Section
Status: Completed | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CAE2C/A
Record Dates: First submitted 2015-09-14; First posted 2015-10-29 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Caesarean Section Born Children
MeSH Terms: interventions — Prebiotics; Probiotics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool samples will be collected from subjects at least once during study visits.
  Voluntary blood sample will be collected from subjects.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Prebiotics group: No intervention since is a follow-up study
  Interventions: Other: Prebiotics
- Prebiotics & Probiotics group: No intervention since is a follow-up study
  Interventions: Other: Prebiotics & Probiotics
- Control group: No intervention since is a follow-up study

INTERVENTIONS:
Other: Prebiotics — To study the long term effect of supplementation in early life
  Groups: Prebiotics group
Other: Prebiotics & Probiotics — To study the long term effect of supplementation in early life
  Groups: Prebiotics & Probiotics group

SUMMARY:
This study investigate the long term effect of supplementation of pre- and probiotics in early life in children born by Caesarean Section.

DETAILED DESCRIPTION:
This is an extension of investigation on the long term effect of supplementation of pre- and probiotics in early life in children born by Caesarean Section from an earlier completed study.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the Julius SN study until 16 weeks of age
* Written informed consent from parent(s) or legally acceptable representatives

Exclusion Criteria:

* Investigator's uncertainty about the willingness or ability of the child and parents to comply with the protocol requirements.

Ages: 36 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who had completed Juliu Sn study until 16 weeks of age.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2015-11; Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Absolute count of Bifidobacterium | 3 - 4 years old
  Difference in absolute count of bifidobacterium between study groups
Absolute level of fecal lactate | 3 - 4 years old
  Difference in absolute level of fecal lactate between study groups
Incidence of allergy manifestation | 3 - 4 years old
  Difference in parent-reported cumulative incidences of allergy manifestation between study groups
Incidence of gastrointestinal symptoms | 3 - 4 years old
  Difference in parent-reported cumulative incidences of gastrointestinal symptoms between study groups
Incidence of infection | 3 - 4 years old
  Difference in parent-reported cumulative incidences of infection between study groups

CONTACTS AND LOCATIONS:
Overall Officials: Mei Chien Chua, Dr, Principal Investigator — KK Women's and Children's Hospital
Locations (2):
- KK Women's and Children's hospital, Singapore, Singapore
- King Chulalongkorn hospital, Bangkok, Thailand